CLINICAL TRIAL: NCT04644588
Title: Correlation Between Scapular Alignment and Upper Limb Function in Children With Hemiparetic Cerebral Palsy
Brief Title: Scapular Alignment and Upper Limb Function in Children With Cerebral Palsy
Acronym: Hemiparesis
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Elsayed Abbass, Dr.Mai Elsayed Abbass, Lecturer of pediatric physical therapy, Cairo University
Other Study IDs: REC\012\002554
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children being assessed for scapular alignment and upper limb function.: Children with hemiparetic cerebral palsy being assessed for scapular alignment and hand function using postural zone software to assess scapular alignment and pediatric arm function test toassess upper limb function .
  Interventions: Diagnostic Test: Children with hemiparetic cerebral palsy being assessed for scapular alignment and upper limb function.

INTERVENTIONS:
Diagnostic Test: Children with hemiparetic cerebral palsy being assessed for scapular alignment and upper limb function. — Children with hemiparetic cerebral palsy being assessed for scapular alignment and upper limb function.
  Other Names: Children being assessed for scapular alignment and upper limb function.

SUMMARY:
Purpose: To determine the effect of scapular alignment on upper limb function in hemiparetic children and to find relation between scapular alignment of the affected, less affected limb and the upper limb function in children with spastic hemiparesis Subjects: Forty children with spastic hemiparetic cerebral palsy, from both genders, were included in this study. They were selected from Outpatient Clinic of Faculty of Physical Therapy, Cairo University. The age of the selected children was ranging from 3 to 6 years old. Degree of spasticity is ranging from 1 to 1+ according to modified Ashworth scale.

Methods: Forty children with spastic hemiparetic cerebral palsy were assessed for scapular alignment using Postural zone software and for upper limb function using pediatric arm function test.

DETAILED DESCRIPTION:
Subjects:

Forty children with spastic hemiplegic CP, from both genders, were included in this study. They were selected from Outpatient Clinic of Faculty of Physical Therapy, Cairo University.

Inclusion criteria:

Children were enrolled in this study according to the following criteria:

1. The age of the selected children was ranging from 3 to 6 years old .
2. Both genders were included.
3. They were able to follow instructions and understand commands.
4. Degree of spasticity is ranging from 1 to 1+ according to modified Ashworth scale.
5. Postural zone software was assess scapular alignment and pediatric arm function test was assess upper arm function .

Exclusion criteria:

The child was excluded from the study if he / she has one or more of the following:

1. Upper limb surgery in the last 12 months.
2. Children which had contracture, fracture, and fixed deformities in the upper limb.
3. Children with muscleoskletal abnormalities as fixed back deformities.

Methods:

Forty children with spastic hemiparetic cerebral palsy were assessed for scapular alignment using Postural zone software and for upper limb function using pediatric arm function test.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the selected children was ranging from 3 to 6 years old .
2. Both genders were included.
3. They were able to follow instructions and understand commands.
4. Degree of spasticity is ranging from 1 to 1+ according to modified Ashworth scale.

Exclusion Criteria:

1. Upper limb surgery in the last 12 months.
2. Children which had contracture, fracture, and fixed deformities in the upper limb.
3. Children with muscleoskletal abnormalities as fixed back deformities.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Forty children with spastic hemiplegic CP, from both genders, were included in this study. They were selected from Outpatient Clinic of Faculty of Physical Therapy, Cairo University.
  The age of the selected children was ranging from 3 to 6 years old. They were able to follow instructions and understand commands.Degree of spasticity is ranging from 1 to 1+ according to modified Ashworth scale.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Number of Children being assessed for scapular alignment. | baseline ( enrolment)
  Children being assessed for scapular alignment using postural zone software.
Number of Children being assessed for upper limb function. | baseline ( enrolment)
  Children being assessed for upper limb function using pediatric arm function test.

CONTACTS AND LOCATIONS:
Overall Officials: Mai Abbass, Ph.D., Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No